CLINICAL TRIAL: NCT06188884
Title: 2018 Classification of Periodontitis Cases: Staging and Grading in Daily Dental Practice of Periodontists, Clinicians With Expertise in Periodontics and General Dental Practitioners
Brief Title: Staging and Grading of Periodontitis: Five Years Later
Status: Not yet recruiting | Type: Observational
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Fabrizio Guerra, Associate professor MED/28, University of Roma La Sapienza
Other Study IDs: NCPD
Record Dates: First submitted 2023-12-18; First posted 2024-01-03 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Periodontal Diseases; Periodontitis
Keywords: periodontitis; classification; periodontal diseases; diagnosis
MeSH Terms: conditions — Periodontal Diseases; Periodontitis; Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to investigate the ability of Periodontists, Clinicians with Expertise in Periodontics and General Dental Practitioners to diagnose periodontitis using the 2017 AAP / EFP World Workshop classification of periodontal diseases.

The purpose of this study is to conduct a online survey in order to:

1. investigate Italian dentists' knowledge on the new classification of periodontal diseases.
2. evaluate the reliability of the diagnosis between different examiners in classifying periodontitis;
3. evaluate the accuracy of the use of grading in the diagnosis of periodontitis;
4. evaluate diagnostic accuracy of staging application in classifying periodontitis.

DETAILED DESCRIPTION:
Four well-documentated clincial cases will be presented to Italian dentists (Periodontists, Clinicians with Expertise in Periodontics and General Dental Practitioners) through online survey to obtain a Clinical application of the 2018 classification of periodontal diseases Each participant will be asked to diagnose periodontitis using staging and grading for each clinical case.

Each periodontal case will be documentated according a previous study (Marini et al. 2022) specifing:

Age; Systemic diseases (presence/absence); Cigarette consumption ( <10 cig/day or >10cig/day); Tooth mobility (presence/absence) Tooth migration (presence/absence) Number of tooth loss due periodontitis (0; <4; > 5) Gingival bleeding (presence/absence) Familiarity for periodontitis

Each periodontal case will be presented showing:

Intra-oral photographs; Full-mouth periapical radiographs; Periodontal chart

ELIGIBILITY:
Inclusion Criteria:

Periodontists, Clinicians With Expertise in Periodontics General Dental Practitioners

Ages: 23 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Periodontists, Clinicians With Expertise in Periodontics General Dental Practitioners
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
evaluate the reliability of the diagnosis between different examiners in classifying periodontitis; | at the moment of the diagnosis
  periodontal diagnosis using I to IV stage and A to C grade.
evaluate diagnostic accuracy of the use of staging in the diagnosis of periodontitis; | at the moment of the diagnosis
  periodontal diagnosis using I to IV stage
evaluate diagnostic accuracy of the use of grading in the diagnosis of periodontitis; | at the moment of the diagnosis
  periodontal diagnosis using A to C grade

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: SAP, CSR
Time Frame: PD and any additional supporting information will become available when summary data are published.
Access Criteria: according to journal policy

REFERENCES:
- [Result] Abrahamian L, Pascual-LaRocca A, Barallat L, Valles C, Herrera D, Sanz M, Nart J, Figuero E. Intra- and inter-examiner reliability in classifying periodontitis according to the 2018 classification of periodontal diseases. J Clin Periodontol. 2022 Aug;49(8):732-739. doi: 10.1111/jcpe.13618. Epub 2022 Jun 22. PMID 35322458
- [Result] Papapanou PN, Sanz M, Buduneli N, Dietrich T, Feres M, Fine DH, Flemmig TF, Garcia R, Giannobile WV, Graziani F, Greenwell H, Herrera D, Kao RT, Kebschull M, Kinane DF, Kirkwood KL, Kocher T, Kornman KS, Kumar PS, Loos BG, Machtei E, Meng H, Mombelli A, Needleman I, Offenbacher S, Seymour GJ, Teles R, Tonetti MS. Periodontitis: Consensus report of workgroup 2 of the 2017 World Workshop on the Classification of Periodontal and Peri-Implant Diseases and Conditions. J Periodontol. 2018 Jun;89 Suppl 1:S173-S182. doi: 10.1002/JPER.17-0721. PMID 29926951
- [Result] Tonetti MS, Greenwell H, Kornman KS. Staging and grading of periodontitis: Framework and proposal of a new classification and case definition. J Periodontol. 2018 Jun;89 Suppl 1:S159-S172. doi: 10.1002/JPER.18-0006. PMID 29926952
- [Result] Marini L, Tonetti MS, Nibali L, Sforza NM, Landi L, Cavalcanti R, Rojas MA, Pilloni A. Implementation of a software application in staging and grading of periodontitis cases. Oral Dis. 2024 Mar;30(2):719-728. doi: 10.1111/odi.14370. Epub 2022 Sep 20. PMID 36083695